CLINICAL TRIAL: NCT06089161
Title: Personalized Obstructive Sleep Apnea Treatment and Effects on Alzheimer's Disease Biomarkers and Cognition Among Blacks
Acronym: PRAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Girardin Jean-Louis, Distinguished Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20220509; 5R01AG075007-02 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Group (Active Comparator): Participants in this group receive the standard of care treatment for sleep apnea for up to six months.
  Interventions: Other: Standard of Care
- Personalized OSA Treatment Group (Experimental): Participants in this group receive personalized OSA treatment for sleep apnea for up to six months.
  Interventions: Other: Standard of Care; Behavioral: Personalized OSA Treatment

INTERVENTIONS:
Other: Standard of Care — Participants in this group will receive standard of care treatment for sleep apnea.
Behavioral: Personalized OSA Treatment — Participants in this group will receive standard of care treatment plus the personalized treatment that consists of videos approximately three minutes long, virtual, accessed through web based application, that the participant watches weekly. The purpose of the video is tailored educational content for sleep apnea.
  Arms: Personalized OSA Treatment Group

SUMMARY:
The purpose of this research is to see how effective the Personalized obstructive sleep apnea (OSA) Treatment Adherence Model called PRAISE is in helping the patient stick to the physician recommended OSA treatment plan Positive Airway Pressure (PAP).

ELIGIBILITY:
Inclusion Criteria:

* Self-reported race/ethnicity as African American, African, Caribbean or black
* Ages 60-85 years
* accessible by phone
* OSA diagnosis
* consent, including permission to release medical data

Exclusion Criteria:

* progressive illnesses in which disability or death is expected within 1 year
* impaired cognitive/ functional ability precluding participation
* intention to move within the year
* and a family member currently enrolled.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants adherence to OSA treatment | Up to 6 months
  The proportion of participants who answer yes (meaning a participant acknowledges an average of more than 4 hours of continuous positive airway pressure use) or no (meaning a participant acknowledges an average of less than 4 hours of continuous positive airway pressure use).

SECONDARY OUTCOMES:
Change in Molecular Biomarkers | Baseline and 6 months
  The molecular biomarker are C₂N, Homocysteine, Neurofilament light, Glial fibrillary acidic protein, Tau, and Amyloid-Beta peptides and the inflammatory markers are Interleukin-6,Interleukin -10, and Tumor Necrosis Factor-alpha. All will be measured in picograms per milliliter.
Change in Vascular Markers | Baseline and 6 months
  Red Blood Cell Count, White Blood Cell Count, and Platelet Count will be measured. All will be measured in Cells/L.
Change in Cardiometabolic Biomarkers measured in mg/dl | Baseline and 6 months
  Total Cholesterol, HDL, LDL, Triglycerides, Bilirubin, Blood Urea Nitrogen (BUN), Calcium, Creatinine, and Glucose. Measured in milligrams/deciliter (mg/dl) assessed with blood analyses.
Change in Cardiometabolic Biomarkers as measured in grams per deciliter | Baseline and 6 months
  Hemoglobin, Albumin, and Total Protein. Measured in grams per deciliter assessed with blood analyses.
Change in Cardiometabolic Biomarkers measured in mmol/mol | Baseline and 6 months
  Glucose/HbA1C, Chloride, Potassium, Sodium, Homocysteine. Measured in mmol/mol assessed with blood analyses
Change in Cardiometabolic Biomarkers- platelet count | Baseline and 6 months
  Platelet Count. Measured per microliter of Blood.
Change in Cardiometabolic Biomarkers as measured per microliter of Blood. | Baseline and 6 months
  Blood Pressure. Measured per microliter of Blood.
Change in Cardiometabolic Biomarkers as measured by Milli-international units per litre. | Baseline and 6 months
  Thyroid-stimulating hormone. Measured Milli-international units per litre.
Change in Cardiometabolic Biomarkers as measured milligrams per liter | Baseline and 6 months
  C-reactive protein Highly Sensitive. Measure milligrams per liter.
Change in Cardiometabolic Biomarkers Measured in microgram | Baseline and 6 months
  Folate. Measured microgram.
Change in Cardiometabolic Biomarkers Measured picograms per milliliter | Baseline and 6 months
  Vitamin B12. Measured picograms per milliliter.
Change in NIH Toolbox -Oral Reading Recognition Test | Baseline, 6 months
  An assessment of reading decoding skills and crystalized abilities. Participants are asked to read aloud letters and words, pronouncing the words as accurately as possible.
Change in NIH Toolbox Picture Vocabulary Test | Baseline, 6 months
  An assessment of receptive vocabulary administered in a computer-adaptive test (CAT) format. Participants must choose which of four pictures best represents a word presented via audio.
Change in NIH Toolbox- Flanker Inhibitory Control and Attention | Baseline, 6 months
  An assessment of inhibitory control and attention. The participant is asked to focus on a particular stimulus while inhibiting attention to the stimuli flanking it. This outcome will be reported as a composite score.
Change in Executive Function measured by Dimensional Change Card Sort Test | Baseline, 6 months
  Executive function, An assessment of cognitive flexibility and attention. The participant is asked to match a series of picture pairs to a target picture.
Change in Episodic memory measured by Picture Sequence Memory Test | Baseline, 6 months
  Episodic memory, An assessment of episodic memory. Participants are shown a number of activities, and then asked to reproduce the sequence of pictures as it was presented.
Change in NIH Toolbox- Auditory Verbal Learning Test | Baseline, 6 months
  Participants are given three trials to recall as many words as possible from a list of fifteen unrelated words. After a 5-25 minute delay, participants are asked to freely recall as many of the 15 words as possible..
Change in Working Memory measured by List Sorting Task | Baseline, 6 months
  Working memory, An assessment of working memory. The participant is asked to recall and sequence different stimuli that are presented visually and via audio.
Change in Processing Speed measured by Patten Comparison Processing Speed Test | Baseline, 6 months
  Processing speed, An assessment of processing speed. Participants are asked to quickly determine whether two stimuli are the same or not the same.
Change in Working Memory measured by Number Span Subset | Baseline, 6 months
  In this test, the participant is asked to recall a series of numbers in reverse order. The correctly recalled series are scored as 1, and the test contains 14 sequences of numbers. The range of working memory score is from 0 to 14, with higher values representing better outcome.
Change in Health-related quality of life | Baseline, 2 months, 6 months
  Patient-Reported Outcomes Measurement Information System Short Form v1.1 - Global Health (5. Excellent, 4. Very good, 3. Good, 2. Fair, 1. Poor) Higher score indicates better self-reported health-related quality of life
Change in Daytime functioning | Baseline, 2 months, 6 months
  Patient-Reported Outcomes Measurement Information System Short form v1.0 Sleep-Related Impairment 8a (1. Not at all 2. A little bit 3. Somewhat 4. Quite a bit 5. Very much) A lower score indicates better daytime functioning
Changes in Sleep Quality measured by Patient-Reported Outcomes Measurement Information System Short Form v1.0 Sleep Disturbance | Baseline, 2 months, 6 months
  Patient-Reported Outcomes Measurement Information System Short Form v1.0 Sleep Disturbance 4a (1. Not at all 2. A little bit 3. Somewhat 4. Quite a bit 5. Very much)
Changes in number of minutes as measured by FitBit Sleep Stages | Baseline, 2 months, 6 months
  Sleep quality will be measured by the number of minutes by FitBit Sleep Stages.
Changes in Sleep quality measured by Sleep Score | Baseline, 2 months, 6 months
  FitBit Sleep score:
  Excellent: 90 to 100 Good: 80 to 89 Fair: 60 to 79 Poor: less than 60 Min: 1 Max: 100 Excellent: 90-100 Good: 80-89 Fair: 60-79 Poor: Less than 60
Change in Cardiometabolic Biomarkers as measured in percentage | Baseline and 6 months
  Hematocrit. Measured as a percentage.
Change in number of calories burned measured by FitBit | Baseline, 2 months, 6 months
  Number of Calories burned
Change in the number of floors climbed measured by Fitbit | Baseline, 2 months
  Number of floors climbed
Change in distance traveled measured in Miles by Fitbit | Baseline, 2 months
  distance traveled measured by mile
Change in number of steps taken measured by Fitbit | Baseline, 2 months
  number of steps taken
Change in Sleep Awakening measured by Fitbit | Baseline, 2 months
  Number of awakenings

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean-Louis, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No